CLINICAL TRIAL: NCT03852251
Title: A Multicenter, Open-label, Phase Ib/II Study of AK104, a PD-1/CTLA-4 Bispecific Antibody, in Subjects With Advanced Solid Tumors or AK104 in Combination With Oxaliplatin and Capecitabine As First-line Therapy in Subjects With Advanced Unresectable or Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma
Brief Title: A Study of AK104, a PD-1/CTLA-4 Bispecific Antibody, for Advanced Solid Tumors or With mXELOX/XELOX as First-line Therapy for Advanced Gastric or GEJ Adenocarcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Collaborators: Akeso Pharmaceuticals, Inc. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AK104-201
Record Dates: First submitted 2019-02-21; First posted 2019-02-25 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Gastric Adenocarcinoma; Advanced Solid Tumors; Gastroesophageal Junction Adenocarcinoma
Keywords: immuno-oncology; PD-1/CTLA-4 Bispecific; gastric or GEJ adenocarcinoma; PD-1; CTLA-4
MeSH Terms: conditions — Diabetes Mellitus, Insulin-Dependent, 12 | interventions — Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AK104 (Experimental): AK104 IV every 2 weeks (q2w)
  Interventions: Biological: AK104
- AK104 and chemotherapy (Experimental): AK104 IV Q2W or Q3W，oxaliplatin IV 85 mg/m2 Q2W or 130mg/m2 Q3W，capecitabine 1000 mg/m2#twice a day (bid) for day 1to day 10 or day 1 to day 14 per cycle
  Interventions: Biological: AK104; Drug: Oxaliplatin; Drug: Capecitabine

INTERVENTIONS:
Biological: AK104 — Subjects will receive AK104 by intravenous administration.
Drug: Oxaliplatin — Subjects will receive AK104 in combination with oxaliplatin and capecitabine.
  Arms: AK104 and chemotherapy
Drug: Capecitabine — Subjects will receive AK104 in combination with oxaliplatin and capecitabine.
  Arms: AK104 and chemotherapy

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics (PK), immunogenicity, pharmacodynamics (PD) and anti-tumor activities of AK104，a PD-1/CTLA-4 bispecific antibody, when administered as a single agent in adults subjects with advanced or metastatic solid tumors, or combined with oxaliplatin and capecitabine as first-line therapy in adult subjects with advanced unresectable or metastatic gastric or gastroesophageal junction (GEJ) adenocarcinoma.

DETAILED DESCRIPTION:
The study consists of a dose escalation and expansion phase (Phase Ib) to determine the recommended Phase 2 dose (RP2D) for AK104 in combination with oxaliplatin and capecitabine, and a dose confirmation phase (Phase II) which will further characterize the treatment of AK104 in combination at the RP2D.

ELIGIBILITY:
Inclusion Criteria:

* Written and signed informed consent.
* Eastern Cooperative Oncology Group (ECOG) Performance Score of 0 or 1.
* Estimated life expectancy of ≥3 months.
* For Phase Ib Cohort 1, histologically or cytologically documented advanced or metastatic solid tumor that is refractory/relapsed to standard therapies, or for which no effective standard therapy is available. For other cohorts in Phase Ib and Phase II, histologically or cytologically documented advanced unresectable or metastatic gastric adenocarcinoma or gastroesophageal Junction (GEJ) adenocarcinoma.
* For cohorts other than cohort 1 in Phase Ib and Phase II: No prior systemic chemotherapy for advanced or metastatic gastric or GEJ adenocarcinoma. Subjects who have received prior adjuvant chemotherapy or neoadjuvant chemotherapy with curative intent, or definitive chemoradiotherapy for advanced disease, will be eligible provided that progression has occurred >6 months from last treatment.
* Subjects must have at least one measurable lesion in accordance with RECIST v1.1. A lesion previously treated with local therapies such as radiotherapy can be considered a target lesion if there is objective evidence of progression in the lesion.
* For cohorts other than cohort 1 in Phase Ib and Phase II: Subjects must provide an available tumor tissue samples taken < 6 months prior to first dose of study treatment.
* Adequate organ function.
* Females of childbearing potential who are sexually active with a nonsterilized male partner must use at least one highly effective method of contraception.
* Nonsterilized males who are sexually active with a female partner of childbearing potential must use highly effective method of contraception from Day 1 and for 120 days after the last dose of investigational product.

Exclusion Criteria:

* Subjects with known HER2-positive gastric or GEJ adenocarcinoma (not applicable for Cohort 1 in Phase Ib).
* Subjects squamous cell, undifferentiated or other histological types of with gastric or GEJ cancer (not applicable for Cohort 1 in Phase Ib).
* Other invasive malignancies within 2 years, except for locally treatable (manifested as cured) malignancies, such as basal or skin squamous cell carcinoma, superficial bladder cancer, cervical or breast carcinoma in situ.
* Receipt of last radiotherapy or any anti-tumor treatment [chemotherapy, targeted therapy, immunotherapy, Chinese patent drugs with antitumor indications, or immunomodulators or tumor embolization] within 4 weeks prior to the first dose of study treatment.
* Prior exposure to any anti-PD-1, anti-PD-L1, anti-CTLA-4 antibody, or any other antibody or drug therapy for T cell co-stimulatory or checkpoint pathways, such as ICOS or agonists (e.g. CD40, CD137, GITR and OX40 etc).
* Subjects with active, known or suspected autoimmune disease, or a medical history of autoimmune disease, with the exceptions of the following: vitiligo, alopecia, Grave disease, psoriasis or eczema not requiring systemic treatment within the last 2 years, hypothyroidism (caused by autoimmune thyroiditis) only requiring steady doses of hormone replacement therapy and type I diabetes only requiring steady doses of insulin replacement therapy, or completely relieved childhood asthma that requires no intervention in adulthood, or primary diseases that will not relapse unless triggered by external factors.
* Active or previously documented inflammatory bowel disease (e.g. Crohn's disease, ulcerative colitis or chronic diarrhea). Inability to swallow, malabsorption syndrome, uncontrollable nausea, vomiting, diarrhea, or other gastrointestinal diseases which significantly affect the absorption of administered drug.
* Known history of primary immunodeficiency virus infection.
* Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
* Known history of interstitial lung disease.
* Known history of active tuberculosis (TB).
* Serious infections within 4 weeks prior to the first dose of study drug, including but not limited to complications requiring hospitalization, sepsis or severe pneumonia.
* An active infection requiring systemic therapy.
* Subjects with untreated chronic hepatitis B or chronic hepatitis B virus (HBV) DNA exceeding 500 IU/ mL or active hepatitis C virus (HCV) should be excluded. Subjects with non-active HBsAg carriers, treated and stable hepatitis B (HBV DNA <500 IU/ mL) , and cured hepatitis C can be enrolled. Subjects with positive HCV antibodies are eligible only if the HCV RNA test results are negative.
* Known history of testing positive for human immunodeficiency virus (HIV).
* Central nervous system (CNS) metastasis, meningeal metastasis, spinal cord compression, or leptomeningeal disease.
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage.
* Clinically active hemoptysis, active diverticulitis, peritoneal abscess, or gastrointestinal obstruction.
* Clinically significant bleeding symptoms or significant bleeding tendency such as gastrointestinal bleeding, hemorrhagic gastric ulcer or vasculitis within 1 month prior to the first dose of study treatment.
* Unresolved toxicities from prior anticancer therapy, defined as having not resolved to NCI CTCAE v5.0 Grade 0 or 1, or to levels dictated in the inclusion/exclusion criteria.
* Receipt of live or attenuated vaccination within 30 days prior to the first dose of study treatment, or plan to receive live or attenuated vaccine during the study.
* Known history of serious hypersensitivity reaction to other monoclonal antibodies.
* Subjects with known contraindications to XELOX（refer to the package inserts of oxaliplatin and capecitabine）(not applicable for Cohort 1 in Phase Ib).
* Known history of allergy or hypersensitivity to AK104 or any of its components (applicable for all cohorts in Phase Ib and Phase II), or oxaliplatin, other platinum compounds, capecitabine, or any of their components (not applicable for Cohort 1 in Phase Ib).
* Any conditions that, in the investigator's opinion, may put subjects treated with the study drug at risks, or interfere with the evaluation of study drug or subject safety, or the interpretation of results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Actual)
Dates: Start 2019-01-18 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2024-03-25 (Actual)

PRIMARY OUTCOMES:
The number of subjects experiencing adverse events (AEs) (Phase Ib) | From the time of informed consent through 90 days following termination of treatment with investigational product
  An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product temporally associated with the use of study treatment, whether or not considered related to the study treatment.
The number of subjects experiencing dose-limiting toxicities (DLTs) (Phase Ib) | During the first 4 weeks
  DLTs will be assessed during the first 4 weeks of treatment for dose-escalation phase and are defined as toxicities that meet pre-defined severity criteria, and assessed as having a suspected relationship to study drug, and unrelated to disease, disease progression, inter-current illness, or concomitant medications that occurs within the first cycle (4 weeks) of treatment.
Anti-tumor activity of AK104 using objective response rate (ORR) based on RECIST v1.1 as assessed by the investigator (Phase II) | From the first dose of study drug through the date of first documented progression, end of study, date of death, or one year after the last patient starts treatment, whichever should occur first
  The ORR is defined as the proportion of subjects with confirmed CR or confirmed PR, based on RECIST Version 1.1.

SECONDARY OUTCOMES:
Disease control rate (DCR) | Up to 2 years
  The DCR is defined as the proportion of subjects with CR, PR, or SD (subjects achieving SD will be included in the DCR if they maintain SD for ≥8 weeks) based on RECIST Version 1.1.
Duration of response (DoR) | Up to 2 years
  Duration of response is defined as the duration from the first documentation of objective response to the first documented disease progression or death due to any cause, whichever occurs first.
Progression-free survival (PFS) | Up to 2 years
  Progression-free survival is defined as the time from the start of treatment with AK104 until the first documentation of disease progression or death due to any cause, whichever occurs first.
Overall survival (OS) | Up to 2 years
  Overall survival is defined as the time from the start of treatment with AK104 until death due to any cause.
Maximum observed concentration (Cmax) of AK104 | From first dose of AK104 through to 90 days after last dose of AK104
  The endpoints for assessment of PK of AK104 include serum concentrations of AK104 at different timepoints after AK104 administration.
Minimum observed concentration (Cmin) of AK104 at steady state | From first dose of AK104 through to 90 days after last dose of AK104
  The endpoints for assessment of PK of AK104 include serum concentrations of AK104 at different timepoints after AK104 administration.
Area under the curve (AUC) of AK104 | From first dose of AK104 through to 90 days after last dose of AK104
  The endpoints for assessment of PK of AK104 include serum concentrations of AK104 at different timepoints after AK104 administration.
Number of subjects who develop detectable anti-drug antibodies (ADAs) | From first dose of AK104 through 90 days after last dose of AK104
  The immunogenicity of AK104 will be assessed by summarizing the number of subjects who develop detectable anti-drug antibodies (ADAs).

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Peng J, Zhu Q, Peng Z, Chen Z, Liu Y, Liu B. Patients with positive HER-2 amplification advanced gastroesophageal junction cancer achieved complete response with combined chemotherapy of AK104/cadonilimab (PD-1/CTLA-4 bispecific): A case report. Front Immunol. 2022 Dec 8;13:1049518. doi: 10.3389/fimmu.2022.1049518. eCollection 2022. PMID 36569905